CLINICAL TRIAL: NCT04561570
Title: Long Term Outcomes of Vivity IOL Versus Control
Brief Title: Long Term Outcomes of Vivity Intra Ocular Lens(IOL) Versus Control
Acronym: REVIVE
Status: Completed | Type: Observational
Sponsor: John Berdahl, MD (Other)
Collaborators: Alcon Research (Industry); The Eye Associates (Other); Eye Care Specialists (Unknown); NewsomeEye (Unknown)
Responsible Party: Sponsor-Investigator, John Berdahl, MD, Principal Investigator, Vance Thompson Vision
Organization: Vance Thompson Vision (Other)
Other Study IDs: The REVIVE Study
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Study Group: Vivity ACRYSOF IQ IOL: Subjects that were implanted with the Vivity ACRYSOF IQ extended depth of focus IntaOcular Lens
  Interventions: Device: Vivity ACRYSOF IQ IOL Group
- Control Group: ACRYSOF IQ IOL: Control Group: Subject that were implanted with the ACRYSOF IQ Monofocal IntaOcular Lens
  Interventions: Device: ACRYSOF IQ IOL Control Group

INTERVENTIONS:
Device: Vivity ACRYSOF IQ IOL Group — Subjects that were implanted with the Vivity ACRYSOF IQ extended depth of focus IntaOcular Lens
  Groups: Study Group: Vivity ACRYSOF IQ IOL
Device: ACRYSOF IQ IOL Control Group — Subject that were implanted with the ACRYSOF IQ Monofocal IntaOcular Lens
  Groups: Control Group: ACRYSOF IQ IOL

SUMMARY:
Evaluate the long-term (>1 yr) outcomes of the Vivity IOL. The investigator will use similar measurements and procedures to the ones performed on these subjects during the FDA clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Must have participated in the FDA study at one of the included sites

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 45-60 subjects will be enrolled (30-45 subjects that received the Vivity IOL and 15-20 subjects that received the control lens in the FDA clinical trial) across up to five investigational sites.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Best Corrected Distance Visual Acuity (BCDVAA) | After 1 year post-op
  Best correct distance visual acuity
Best Corrected Intermediate Visual Acuity (BCIVA) | After 1 year post-op
  Best correct intermediate visual acuity
Defocus Curve | After 1 year post-op

SECONDARY OUTCOMES:
Uncorrected Distance Visual Acuity (UCDVA) | After 1 year post-op
  Uncorrected Distance Visual Acuity
UCNVA | After 1 year post-op
  Uncorrected Near Visual Acuity
Dyphotopsia rate | After 1 year post-op
  Demonstrated by responses on questionnaire
Post-operative IOLSAT | After 1 year post-op
  Questionnaire about satisfaction with your vision after surgery. 0-4 scale with 4 being the worse outcome
(Post-operative QUVID) | After 1 year post-op
  Questionnaire about the quality of your vision after surgery.0-4 scale with 4 being the worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States